CLINICAL TRIAL: NCT04730024
Title: Long-term Follow-up Study to Evaluate the Safety and Explore the Efficacy of Multiple Doses of FURESTEM-AD Inj. for Moderate to Severe Chronic Atopic Dermatitis: 5-year Results From the K0104 Extension Study
Brief Title: Long-term Follow-up Study to Evaluate the Safety and Explore the Efficacy of Multiple Doses of FURESTEM-AD Inj
Status: Not yet recruiting | Type: Observational
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: K0104-E
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Not applicable(observational study) — Not applicable(observational study)

SUMMARY:
A multi-center, open, long-term follow-up study to Evaluate the Safety and Explore the Efficacy of Multiple Doses of FURESTEM-AD inj. for Moderate to Severe Chronic Atopic Dermatitis: 5-year Results from the K0104 Extension Study

ELIGIBILITY:
Inclusion Criteria:

1. Subject who enrolled K0104 Clinical Trial(parent study).
2. Subjects who understand and voluntarily sign an informed consent form

Exclusion Criteria:

1. Subjects who are expected to be unable to perform at least one follow-up during this study (K0104-E)
2. Subjects who has received/administered clinical trial drugs or medical devices by participating in other clinical trials until the first visit of this trial (K0104-E) after the completion of K0104 clinical trial
3. Subjects who are judged to be unsuitable for other researchers to participate in the research

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study (K0104-E), it was planned to select subjects who participated in the K0104 clinical trial, a parent study.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-03-27 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment (Rate of Adverse Event, Number of Participants with Adverse Event) | for 5 years

SECONDARY OUTCOMES:
Percentage of subjects whose EASI decreased by 50% or more at each evaluation visit compared to the baseline (EASI-50) | for 5 years
Percentage of subjects whose Eczema Area and Severity Index (EASI) was decreased from baseline by more than 75% at each visit (EASI-75) | for 5 years
Rate of change and Change in EASI from baseline | for 5 years
  EASI range is from 0 (clear) to 72 (severe)
Percentage of subjects whose Investigator's Global Assessment (IGA) score at each visit is 0 or 1 | for 5 years
Percentage of subjects whose IGA at each visit is 0 or 1, or improved to 2 or higher | for 5 years
Percentage of subjects whose SCORing Atopic Dermatitis (SCORAD) INDEX was decreased from baseline by more than 50% at each visit (SCORAD-50) | for 5 years
Rate of change and Change in SCORAD index from baseline at each visit | for 5 years
  SCORAD index range is from 0 (clear) to 103 (severe)
Change and rate of change in Body Surface Area (BSA) | for 5 years
Change and rate of change in total serum Immunoglobulin E (IgE) | for 5 years
Change and rate of change DLQI | for 5 years
Change and rate of change POEM | for 5 years
Change and rate of change Peak Pruritus NRS | for 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Medical Center, Ilsan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided